CLINICAL TRIAL: NCT06197880
Title: Three-dimensional Evaluation of the Airway Morphology After En-masse Retraction in Bimaxillary Protrusion Patients by Using Cone Beam Computed Tomography
Brief Title: Airway Morphology After En-masse Retraction in Bimaxillary Protrusion Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Rehab Abd El Razek Abd El Aziz Khalil, Lecturer of Orthodontics, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: # REC-FDBSU/07072022-01/AR
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Airway
Keywords: en-masse retraction airway morphology CBCT

STUDY DESIGN:
Intervention Model Description: single-arm clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bimaxillary protrusion (Experimental): En masse retraction
  Interventions: Other: Anterior teeth retraction

INTERVENTIONS:
Other: Anterior teeth retraction — En masse retraction of the upper and lower anterior segments using maximum anchorage

SUMMARY:
This study aims to three-dimensionally assess the changes in the airway morphology after anterior segment retraction using maximum anchorage.

DETAILED DESCRIPTION:
Participants were recruited from the Faculty of Dentistry, Beni-Suef University. All subjects were informed of the treatment procedures and signed a consent form.

Methodology:

The patients were treated by using fixed appliance and extraction of four first premolars. Maximum anchorage was obtained by using miniscrews that were inserted between the maxillary first molars and second premolars. En masse retraction of the upper and lower anterior segments was carried out by using NiTi closed coil springs.

Cone beam computed tomography (CBCT) will be obtained before (T0) and after en masse retraction (T1). CBCT will be used for three-dimensional evaluation of the changes of the airway morphology after en masse retraction of the upper and lower anterior segments with maximum anchorage.

The results will be obtained and statistically evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Class I bimaxillary protrusion requiring extraction of four first premolars and en masse retraction of the anterior segments.
2. Age: 18 - 35 years old.
3. Fair oral hygiene.

Exclusion Criteria:

1. Active periodontal disease.
2. Systemic diseases or medications that alter bone metabolism.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
assess the changes in the airway morphology | 6 months
  measure the airway volume before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Khalil, Principal Investigator — Faculty of Dentistry Beni Suef University
Locations (1):
- Faculty of Dentistry Beni Suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valiathan M, El H, Hans MG, Palomo MJ. Effects of extraction versus non-extraction treatment on oropharyngeal airway volume. Angle Orthod. 2010 Nov;80(6):1068-74. doi: 10.2319/010810-19.1. PMID 20677956
- [Background] Wang Q, Jia P, Anderson NK, Wang L, Lin J. Changes of pharyngeal airway size and hyoid bone position following orthodontic treatment of Class I bimaxillary protrusion. Angle Orthod. 2012 Jan;82(1):115-21. doi: 10.2319/011011-13.1. Epub 2011 Jul 27. PMID 21793712
- [Background] Chen Y, Hong L, Wang CL, Zhang SJ, Cao C, Wei F, Lv T, Zhang F, Liu DX. Effect of large incisor retraction on upper airway morphology in adult bimaxillary protrusion patients. Angle Orthod. 2012 Nov;82(6):964-70. doi: 10.2319/110211-675.1. Epub 2012 Mar 30. PMID 22462464